CLINICAL TRIAL: NCT02188329
Title: National Survey of Early Care and Education
Acronym: NSECE
Status: Completed | Type: Observational
Sponsor: National Opinion Research Center (Other)
Collaborators: Office of Planning, Research & Evaluation (U.S. Federal Agency); Chapin Hall at the University of Chicago (Other); Child Trends (Other); Impaq Intl. (Unknown)
Responsible Party: Principal Investigator, Rupa Datta, Vice President and Senior Fellow, National Opinion Research Center
Other Study IDs: HHHSP23320095647WC, 23337017T
Record Dates: First submitted 2014-02-21; First posted 2014-07-11 (Estimated); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Supply and Demand of Early Care and Education in the US
Keywords: Early care and education; ECE; workforce; child care; caregivers; home-based providers; center-based providers

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Households with children under 13: Interviews were conducted with the parent or guardian of a child or children under age 13.
- Home-based providers: Individuals who provide care in a home-based setting to children under age 13 who are not their own.
- Center-based providers: Directors of early care and education programs that provide care to children not yet in kindergarten.
- Center-based workforce: Classroom-assigned instructional staff sampled from each center-based provider who completed an interview.

SUMMARY:
The primary purpose of the National Survey of Early Care and Education (NSECE) was to provide a comprehensive snapshot of both the availability and utilization of early care and education in the United States. The main objectives of the study included:

* Providing the first national portrait of the availability of early care and education for the full spectrum of care providers, including householders and providers from all 50 states and the District of Columbia.
* Identifying early care and education and school-age care (ECE/SA) needs and preferences among households in the United States with children under age 13 as they pertain to supporting both the employment of parents and the development of children.
* Capturing data on all forms of non-parental care for all children in a household.
* Providing the perspectives of both families and providers on the services offered in a system where children are often in multiple arrangements and providers receive funding from multiple sources.
* Linking the data set collected with policy-relevant data.
* Increasing the understanding of the care received by low-income children and how that varies across communities.

The NSECE is a set of four integrated, nationally representative surveys conducted in 2012. These were surveys of 1) households with children under 13, 2) home-based providers 3) center-based providers, and 4) the center-based provider workforce. Together they characterize the supply of and demand for early care and education in America and permit better understanding of how well families' needs and preferences coordinate with providers' offerings and constraints.

DETAILED DESCRIPTION:
In order to create a comprehensive portrait of the availability and use of early care and education, the NSECE fielded a set of four integrated, nationally representative surveys in 2012. These were surveys of 1) households with children under 13, 2) home-based providers 3) center-based providers, and 4) the center-based provider workforce. Together they characterize the supply of and demand for early care and education in America and permit better understanding of how well families' needs and preferences coordinate with providers' offerings and constraints.

The Household Survey was conducted with a parent or guardian of a child or children under age 13 in households with at least one member child under age 13. Eligible respondents were identified through the Household Screener based only on the presence of an age-eligible child. Screening was completed by mail, by phone, and in person. This survey documents the nation's demand for early care and education services. Key questionnaire topics include details on usage of non-parental care, expenditures on non-parental care, parental search behavior for early care and education, and the balance of parental employment with child care needs and availability. These data will help to answer such research questions as 1) Who is caring for America's children when they are not with their parents and do families with different demographic characteristics have different preferences or different patterns of usage? 2) How do families search for care and how does this vary by age of children, characteristics of parents, location, and availability of licensed slots per population? 3) How and how much do families pay for care? and 4) How many families of different characteristics receive public financial support for ECE, and how does this vary by age of child and type of care utilized?

The Home-Based Provider Survey was conducted with individuals who provide care in a home-based setting for children under age 13 who are not their own. Two sample sources contributed providers. One, home-based providers who appeared in provider sampling frames constructed from state and national lists were sampled for this survey. We designated these providers as 'listed.' Listed providers were primarily licensed or regulated family day care providers, but also included other formally listed home-based providers such as license-exempt providers or providers participating in Early Head Start. Alternatively, households could have been identified as eligible based on their responses to the household screener (specifically, that an adult in the household regularly cared for children not his or her own at least five hours per week in a home-based setting). These providers did not appear in the provider sampling frame and are designated as 'unlisted.' Data collection was conducted by Internet, in person, and by telephone with field interviewers.

Key questionnaire topics in the home-based provider questionnaire include enrollment and the characteristics of the children served, rates charged for care, participation in government programs, household composition, qualifications for and attitudes toward early childhood education, use of curricula and activities conducted with children (varied to be appropriate for younger children and school-age children). Portions of the home-based provider questionnaire will contribute to analyses of the ECE workforce and mirror the content of the workforce questionnaire administered to classroom-assigned instructional staff at center-based providers. Other portions of this questionnaire closely mimic the center-based provider questionnaire (see below), so that enrollment, program participation, provider charges for care, attitudes, orientation and activities data can be accurately compared across all different categories of provider. These data will answer such questions as 1) What kind of early care and education is available across communities throughout the country? 2) How well does the available supply of early care and education support parents' employment? 3) How do different types of providers vary in their characteristics of care and affordability? and 4) Who are the individuals working in early care and education? What are their experiences in terms of employment characteristics, classroom activities, and professional development? What are their attitudes, orientations, and stress and depression levels?

The inclusion of providers identified through the Household Screener offers unprecedented nationally representative data on family, friend and neighbor providers and is one of the pioneering aspects of the NSECE. We will learn about both paid and unpaid care, including how they differ in their characteristics and their availability to families.

The Center-Based Provider Survey was conducted with directors of ECE programs that provide care to children not yet in kindergarten who were identified from the provider sampling frame built from state or national administrative lists such as state licensing lists, Head Start program records, or pre-K rolls. These providers included regulated, licensed, and other private providers as well. The center-based provider questionnaire was preceded by a Center-Based Provider Screener that confirmed and updated information from the provider sampling frame, determined the availability of school-age after-school care at elementary schools, and determined eligibility for the center-based provider questionnaire. Topics covered by this instrument include enrollment and characteristics of children served, staffing, prices charged, schedules of service, participation in government programs, and staff compensation and professional development policies. The questionnaire also includes the selection of a representative classroom about which more detailed staffing, compensation, and curriculum information are collected. These data constitute a nationally representative sample of ECE classrooms.

The center-based provider questionnaire data will answer such questions as 1) What kind of early care and education is available across communities throughout the country? 2) How well does the available supply of early care and education support parents' employment? 3) How do different types of providers vary in their characteristics of care and affordability? and 4) How many and what types of providers participate in quality improvement efforts such as staff quality ratings and professional development?

The Workforce Provider Survey sample comprised one classroom-assigned instructional staff person from each center-based provider who completed a center-based provider interview. Workforce respondents were drawn from the center-based provider questionnaire data, in which all staff members had been enumerated from a randomly selected classroom. The questionnaire closely mirrors portions of the home-based provider questionnaire, so that the two data sources together can paint a rich portrait of the paid ECE workforce, including center-based and home-based paid providers. (Individuals who were not paid will be profiled as described in the family, friends, and neighbor section above.) Topics include information about the work setting (activities in the classroom, interactions with parents and other staff, availability of professional development and other supports), roles and responsibilities (lead teacher, teacher, assistant teacher, aide), compensation (wages and benefits), and perceived leadership and morale, as well as personal information about qualifications, attitudes toward ECE, and stress, depression, and demographic information.

The workforce questionnaire is the simplest of the NSECE survey instruments, but these data represent a signal contribution of the study. No nationally representative survey of paid ECE workers has ever been done, yet many of the pressing ECE policy questions require better understanding of home-based care providers' qualifications, access to professional development, motivation for working in the field, and nature of participation in the labor market as well as the extent to which paid home-based providers are more generally available for expanding and improving overall ECE supply. Some of the workforce questionnaire data will allow tabulation by provider program characteristics (such as enrollment size, type of care, geographic location, for-profit/not-for profit status, and participation in government programs) of factors that have been found in the literature to predict observed quality. These factors include staff qualifications and compensation, use of curricula, availability of professional development, and children's activities while in care. The data will answer such questions as who are the individuals working in early care and education and what are their experiences in terms of employment characteristics, classroom activities, and professional development?

ELIGIBILITY:
Inclusion Criteria:

* Households with at least one child under the age of 13.
* Individuals who care for a child under 13 who is not their own in a home- based setting for at least five hours a week.
* Center-based ECE programs that provide care to children not yet in kindergarten who were identified from the provider sampling frame built from state or national administrative lists such as state licensing lists.
* Respondents for the center-based workforce survey are selected from the list of instructional staff associated with the randomly selected classroom from the center-based provider interview.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Households with children under 13 years. Individuals providing at least 5 hours' weekly care to children under 13 years not their own in a home-based setting. Early care and education centers serving children not yet in kindergarten. Individuals working in center-based classrooms.
Sampling Method: Probability Sample
Enrollment: 31436 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Need for and use of childcare in households with children under 13 | At time of interview
  The household questionnaire collected information on each household's need for and use of early care and education services, including details on usage of non-parental care, expenditures on non-parental care, parental search behavior for early care and education, and the balance of parental employment with child care needs and availability.

SECONDARY OUTCOMES:
Provision and characteristics of child care among center-based providers | At time of interview
  The center-based provider questionnaire collected information on enrollment and characteristics of children served, staffing, prices charged, schedules of service, participation in government programs, and staff compensation and professional development policies. The questionnaire also includes the selection of a representative classroom about which more detailed staffing, compensation, and curriculum information are collected.

OTHER OUTCOMES:
Provision and characteristics of child care among home-based providers | At time of interview
  The home-based provider questionnaire collected information on enrollment and the characteristics of the children served, rates charged for care, participation in government programs, household composition, qualifications for and attitudes toward early childhood education, use of curricula and activities conducted with children (varied to be appropriate for younger children and school-age children). Portions of the home-based provider questionnaire will contribute to analyses of the ECE workforce and mirror the content of the workforce questionnaire administered to classroom-assigned instructional staff at center-based providers.
Characteristics and experiences of the ECE workforce | At the time of interview
  The workforce questionnaire collected information about the work setting (activities in the classroom, interactions with parents and other staff, availability of professional development and other supports), roles and responsibilities (lead teacher, teacher, assistant teacher, aide), compensation (wages and benefits), and perceived leadership and morale, as well as personal information about qualifications, attitudes toward ECE, and stress, depression, and demographic information.

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Goerge, PhD, Principal Investigator — Chapin Hall at the University of Chicago
Locations (1):
- NORC at the University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] National Survey of Early Care and Education Project Team. (2013). National Survey of Early Care and Education: Summary Data Collection and Sampling Methodology. OPRE Report #2013-46, Washington DC: Office of Planning, Research and Evaluation, Administration for Children and Families, U.S. Department of Health and Human Services.